CLINICAL TRIAL: NCT06006130
Title: Investigating the Neurobiological Contributions to Pain in Patients With Fibromyalgia
Brief Title: Neurophysiology of Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16482
Record Dates: First submitted 2023-07-28; First posted 2023-08-23 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; transcranial magnetic stimulation; neuroplasticity; pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Experiment 1: Response to real intervention compared between fibromyalgia and healthy control group Experiment 2: Fibromyalgia participants allocated to real or sham intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: Experiment 1: Outcomes assessor will be blinded to the groups (fibromyalgia vs controls) the data is obtained from Experiment 2: Outcomes assessor and participants will be blinded to the intervention group that participants are allocated to (sham vs real treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Active Comparator): Repetitive Transcranial Magnetic Stimulation (rTMS) will be delivered at 10 Hz, 1500 pulses targeting the hand representation of the left primary motor cortex. rTMS delivery will require ~11 min to complete. In Experiment 1, this intervention will be performed for 1 session (~11min). In Experiment 2, this intervention will be performed approximately 5 days per week for 2 weeks. In addition, participants will experience their standard medical care.
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): Sham rTMS will be delivered at as a placebo control. It is important to note that from the participant perspective, the sham stimulation will feel and sound identical to active rTMS. In Experiment 2, this intervention will be performed approximately 5 days per week for 2 weeks. In addition, participants will experience their standard medical care.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a non-invasive, non-painful procedure used to relieve chronic pain and promote short-term changes. The abductor pollicis brevis (APB) muscle of the left motor cortex will be targeted using neuronavigation software. 1500 pulses will be delivered at 10 Hz stimulation. Stimulation will be delivered at 80% of the resting motor threshold obtained from the right APB muscle. The delivery of rTMS requires 11 minutes in total.
  Arms: Active rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — A sham coil will be utilized for the sham rTMS condition. It is important to note that from the participant perspective, the sham stimulation will feel and sound identical to active. The location and all other parameters of Sham rTMS will be identical to Active rTMS.
  Arms: Sham rTMS

SUMMARY:
Fibromyalgia is a syndrome associated with fatigue and chronic pain, leading to significant physical limitations and impaired quality of life. There are several challenges that complicate the diagnosis and management of fibromyalgia. The etiology is not well defined, as there are several proposed factors that may trigger the genesis of pain in fibromyalgia including physical and/or emotional life stressors, and genetic predispositions involving neuromodulator pathways. Chronic pain in fibromyalgia arises in the absence of tissue pathology, and consequently a lack of consensus on reliable diagnostic criteria. Understanding the neurophysiology of fibromyalgia would aid in the discovery of objective biomarkers for diagnosis. Therefore, the goals of this study are to:

1. Compare the neurophysiological responses in fibromyalgia compared to healthy controls.
2. Determine whether a two-week rTMS protocol will alter pain in individuals with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a syndrome associated with fatigue and chronic pain, leading to significant physical limitations and impaired quality of life. Fibromyalgia affects 1.7% of Canadians, with a higher prevalence in females compared to males at 9:1 [1]. There are several challenges that complicate the diagnosis and management of fibromyalgia. The etiology is not well defined, as there are several proposed factors that may trigger the genesis of pain in fibromyalgia. Chronic pain in fibromyalgia arises in the absence of tissue pathology, and consequently a lack of consensus on reliable diagnostic criteria. Understanding the pathophysiology of fibromyalgia would aid in the identification of objective biomarkers that could be used for diagnosis.

Multiple theories have been posited to explain the genesis of chronic pain. The gate control theory describes the attenuation of pain signals in the spinal cord prior to cortical processing, and it has been hypothesized that loss of this gate control leads to the genesis of chronic pain [2]. Gate control can be observed by reduction of afferent signals during active muscle contraction. For example, the amplitude of the somatosensory-evoked potential (SEP) is attenuated during active contraction [3]. To our knowledge, it is unknown whether such gate control is observed in fibromyalgia. The lack of gate control may contribute to chronic pain in this population.

The sensorimotor theory suggests that incongruency between motor intention and sensory feedback underlies chronic pain where there is an absence of tissue pathology [4]. This may align with the genesis of fibromyalgia, given the findings that those with fibromyalgia have altered tactile and proprioceptive functioning [5]. Corticomuscular coherence (CMC) is a useful tool that uses electroencephalography (EEG) and electromyography (EMG) to probe the synchrony of neural firing between the brain and muscle [6]. To our knowledge, it is unknown how the magnitude of CMC varies in fibromyalgia compared to healthy controls.

Non-invasive brain stimulation in the form of Transcranial Magnetic Stimulation (TMS) has been used to probe the activity of corticospinal and cortical networks in fibromyalgia. When TMS pulses are delivered in a repetitive train, a protocol known as repetitive TMS (rTMS), short-term neuroplasticity can be induced (i.e., a change in the activity of neurons in the brain). In fibromyalgia, Mhalla et al. [7] found that 5 days of 10 Hz rTMS reduced pain intensity and improved quality of life metrics. It is unknown whether a longer intervention period could lead to greater analgesic effects.

Finally, central sensitization may explain the widespread chronic pain experienced in fibromyalgia. There are several neuromodulators that contribute to the neurobiology of central sensitization and may be implicated in this condition including serotonin, dopamine, and brain-derived neurotrophic factor (BDNF). Serotonin is linked to pain modulation, such that increased levels of 5-HT are associated with hyperalgesia [8]. BDNF has been implicated in the genesis of neuropathic pain [9]. In fibromyalgia compared to healthy controls, serum BDNF levels have been reported to be higher [10]. Abnormal dopamine function may also be associated with fibromyalgia [11]. Positron-emission tomography (PET) studies show lower cortical dopamine D2/D3 binding availability in fibromyalgia compared to healthy controls [12].

Ultimately, a combination of events may lead to widespread chronic pain in fibromyalgia. Understanding the neurophysiology of fibromyalgia would aid in the discovery of objective biomarkers for diagnosis. Therefore, the goals of this study are to:

1. Compare the neurophysiological responses in fibromyalgia compared to healthy controls.

2. Determine whether a two-week rTMS protocol will alter pain in individuals with fibromyalgia.

1. M. B. Yunus, "The role of gender in fibromyalgia syndrome," Curr Rheumatol Rep, vol. 3, no. 2, pp. 128-134, 2001, doi: 10.1007/S11926-001-0008-3.
2. R. Melzack, "Evolution of the neuromatrix theory of pain. The Prithvi Raj Lecture: presented at the third World Congress of World Institute of Pain, Barcelona 2004," Pain Pract, vol. 5, no. 2, pp. 85-94, Jun. 2005, doi: 10.1111/J.1533-2500.2005.05203.X.
3. H. Nakata, K. Inui, T. Wasaka, Y. Nishihira, and R. Kakigi, "Mechanisms of differences in gating effects on short-and long-latency somatosensory evoked potentials relating to movement," Brain Topogr, vol. 15, no. 4, pp. 211-222, Jun. 2003, doi: 10.1023/A:1023908707851.
4. A. D. Vittersø, M. Halicka, G. Buckingham, M. J. Proulx, and J. H. Bultitude, "The sensorimotor theory of pathological pain revisited," Neurosci Biobehav Rev, vol. 139, Aug. 2022, doi: 10.1016/J.NEUBIOREV.2022.104735.
5. S. Toprak Celenay, O. Mete, O. Coban, D. Oskay, and S. Erten, "Trunk position sense, postural stability, and spine posture in fibromyalgia," Rheumatol Int, vol. 39, no. 12, pp. 2087-2094, Dec. 2019, doi: 10.1007/S00296-019-04399-1/TABLES/2.
6. A. Chowdhury, H. Raza, Y. K. Meena, A. Dutta, and G. Prasad, "An EEG-EMG correlation-based brain-computer interface for hand orthosis supported neuro-rehabilitation," J Neurosci Methods, vol. 312, pp. 1-11, Jan. 2019, doi: 10.1016/J.JNEUMETH.2018.11.010.
7. A. Mhalla et al., "Long-term maintenance of the analgesic effects of transcranial magnetic stimulation in fibromyalgia," Pain, vol. 152, no. 7, pp. 1478-1485, 2011, doi: 10.1016/J.PAIN.2011.01.034.
8. E. A. Ovrom, K. A. ; Mostert, S. ; Khakhkhar, D. P. ; Mckee, P. ; Yang, and Y. F. A. Her, "A Comprehensive Review of the Genetic and Epigenetic Contributions to the Development of Fibromyalgia," Biomedicines 2023, Vol. 11, Page 1119, vol. 11, no. 4, p. 1119, Apr. 2023, doi: 10.3390/BIOMEDICINES11041119.
9. K. Obata and K. Noguchi, "BDNF in sensory neurons and chronic pain," Neurosci Res, vol. 55, no. 1, pp. 1-10, May 2006, doi: 10.1016/J.NEURES.2006.01.005.
10. A. Deitos et al., "Clinical Value of Serum Neuroplasticity Mediators in Identifying the Central Sensitivity Syndrome in Patients With Chronic Pain With and Without Structural Pathology," Clin J Pain, vol. 31, no. 11, pp. 959-967, 2015, doi: 10.1097/AJP.0000000000000194.
11. P. B. Wood, M. F. Glabus, R. Simpson, and J. C. Patterson, "Changes in gray matter density in fibromyalgia: correlation with dopamine metabolism," J Pain, vol. 10, no. 6, pp. 609-618, Jun. 2009, doi: 10.1016/J.JPAIN.2008.12.008.
12. D. S. Albrecht et al., "Differential dopamine function in fibromyalgia," Brain Imaging Behav, vol. 10, no. 3, pp. 829-839, Sep. 2016, doi: 10.1007/S11682-015-9459-4/FIGURES/4.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old

Exclusion Criteria:

* contraindications to TMS
* chronic pain associated with diagnoses other than fibromyalgia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS-29 v2.0 Profile | Experiment 1: At baseline pre-intervention, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  Using numerical rating (0 to 5) to assess the change in seven health domains including physical function, anxiety, depression, fatigue, sleep disturbances, ability to participate in social roles and activities, and pain interference. Each category consists of 4 questions. Also uses a numerical rating to asses pain intensity (0-10).
Change in Fibromyalgia impact questionnaire (FIQ) | Experiment 1: At baseline pre-intervention, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  This instrument will be used to assess the patients feeling and emotion related to their pain experience.

SECONDARY OUTCOMES:
Change in Pain catastrophizing scale-EN-SF | Experiment 1: At baseline pre-intervention, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  Will be used to assess the patients feeling and emotion related to their pain experience
Change in Patient Health Questionnaire-4 (PHQ-4) | Experiment 1: At baseline pre-intervention, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  Will be used to assess for symptoms of for Major Depressive Disorder and Generalized Anxiety Disorder
Change in Short-form Posttraumatic Checklist-5 (Short-form PCL-5) | Experiment 1: At baseline pre-intervention, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  Will be used to screen for symptoms of Posttraumatic Stress Disorder (PTSD)
Change in Motor-evoked potentials (MEPs) | Experiment 1: At baseline pre-intervention and immediately following 1 treatment session, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  This will include an assessments of MEPs obtained using Transcranial Magnetic Stimulation (TMS).
Change in Short-Interval Intracortical Inhibition (SICI) | Experiment 1: At baseline pre-intervention and immediately following 1 treatment session, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  This will include an assessments of SICI obtained using Transcranial Magnetic Stimulation (TMS).
Change in performance on sensorimotor tasks | Experiment 1: At baseline pre-intervention, Experiment 2: At baseline pre-intervention and 2 weeks post-intervention
  Tasks include tactile localization, temporal order judgement (TOJ), and sequential amplitude discrimination
EEG assessment of Somatosensory-evoked potentials (SEPs) | Experiment 1: At baseline pre-intervention only
  This will include an assessment of SEPs using EEG electrodes.
EEG assessment of Pain-related evoked potentials (PREPs) | Experiment 1: At baseline pre-intervention only
  This will include an assessment of PREPs using EEG electrodes.
EEG assessment of Corticomuscular coherence (CMC) | Experiment 1: At baseline pre-intervention only
  This will include an assessment of CMC using EEG electrodes.
EEG assessment of Event-related desynchronization (ERD) | Experiment 1: At baseline pre-intervention only
  This will include an assessment of ERD using EEG electrodes.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No